CLINICAL TRIAL: NCT03872739
Title: To Compare Intravenous and Oral Hydration of the Prevention for Contrast-induced Nephropathy in Elderly Patients Undergoing Intravenous Contrast-enhanced Computed Tomography： A Multi-center Randomized Control Trail
Brief Title: To Compare Intravenous and Oral Hydration of the Prevention for CIN in Elderly Patients Undergoing Intravenous CECT
Acronym: CINOECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yu Danqing (Other)
Responsible Party: Sponsor-Investigator, Yu Danqing, Director,Clinical Professor, Guangdong Academy of Medical Sciences
Organization: Guangdong Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201704020124
Record Dates: First submitted 2019-02-27; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: CIN
Keywords: CIN; Hydration; enhanced computed tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- distilled water (Experimental): Oral distilled water at the rate of 3 mL/kg/h rate during undergoing enhanced computed tomography examination before 1-2 and after 4-6 hours
  Interventions: Procedure: enhanced computed tomography
- Saline (Placebo Comparator): intravenous saline hydration at the rate of 1 mL/kg/h rate during undergoing enhanced computed tomography examination before and after 12 hours
  Interventions: Procedure: enhanced computed tomography

INTERVENTIONS:
Procedure: enhanced computed tomography — undergoing enhanced computed tomography

SUMMARY:
To Compare Intravenous and Oral Hydration of the Prevention for Contrast-induced Nephropathy in Elderly Patients Undergoing Intravenous Contrast-enhanced Computed Tomography.

DETAILED DESCRIPTION:
The prospective multicenter randomized controlled clinical research discusses the comparison of oral and intravenous hydration for prevention of contrast-induced nephropathy in elderly patients with enhanced computed tomography, establishing a simple hydration proposal.

ELIGIBILITY:
Inclusion Criteria:

* Age>21
* informed consent
* Undergoing Intravenous Contrast-enhanced Computed Tomography

Exclusion Criteria:

* CT enhancement was not performed;
* Dialysis treatment of patients with end-stage renal failure or heart, kidney transplantation;
* Exposure to radioactive contrast medium within 48 hours prior to or within 72 hours of examination;
* Acute decompensated heart failure;
* Allergic to radioactive contrast agent;
* Be subjected to life - threatening trauma;
* Severe infection;
* Surgery was performed within 2 days of CT examination.
* Combined with multiple myeloma, urinary obstruction, aortic dissection
* Can cause acute kidney injury disease;
* Use of aminoglycosides and other nephrotoxic drugs 2 weeks before.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1368 (Estimated)
Dates: Start 2016-10-08 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
CIN | 72hours
  Compared with before examination, the increase of serum creatinine conforms to the diagnostic criteria of contrast induced nephropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Danqing Yu, Doctor, Principal Investigator — Guangdong Cardiovascular Institute
Locations (1):
- Guangdong provincial people's hospital, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No